CLINICAL TRIAL: NCT02314624
Title: PracticeGround: Transforming Training and Delivery of Mental Health EBPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evidence-Based Practice Institute, Seattle, WA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2R44MH093993-02A1 (NIH)
Record Dates: First submitted 2014-12-05; First posted 2014-12-11 (Estimated); Results first posted 2023-06-15 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Depression; Insomnia; Suicide
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders; Suicide | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WILLOW (Experimental): Clinicians have access to WILLOW's dynamic progress monitoring, clinical decision support, rich visual displays of client outcomes, online training modules in ESTs, just-in-time training for guided real-time assistance in delivering ESTs, educational videos, and a client portal
  Interventions: Behavioral: Behavioral Activation for Depression, Cognitive Behavior Therapy for Insomnia, Collaborative Assessment and Management of Suicidality
- Treatment-as-Usual (Active Comparator): Usual care without access to WILLOW.
  Interventions: Behavioral: Care-as-Usual Psychotherapy

INTERVENTIONS:
Behavioral: Behavioral Activation for Depression, Cognitive Behavior Therapy for Insomnia, Collaborative Assessment and Management of Suicidality — Evidence-based interventions for treating depression and concurrent problems
  Arms: WILLOW
Behavioral: Care-as-Usual Psychotherapy — Usual care psychotherapy for depression and concurrent problems
  Arms: Treatment-as-Usual

SUMMARY:
The ultimate goal is to facilitate the delivery of empirically supported treatments (ESTs) for mental disorders and to improve client mental health outcomes. Toward this end, this Phase II SBIR proposal seeks to complete the development and testing of PracticeGround, a comprehensive software system designed to integrate with electronic health records, and that contains multiple methods of training clinicians in ESTs and delivering ESTs to clients, continuous progress monitoring of client outcomes, and clinical support tools to guide clinicians and clients through delivery of the necessary EST. The investigators will conduct an 18-week randomized controlled trial (N=80) comparing PracticeGround (n=40) to care-as-usual (n=40) in depressed outpatient clients. PracticeGround clinicians will have full access to the software. Study clinicians and clients will be assessed once every six weeks (baseline, 6, 12, and 18 weeks). To ensure generalizability of findings, the investigators will not control for natural therapy variations (e.g.,session frequency, medication use, etc.). Primary outcomes include: depression, psychological distress, treatment satisfaction (clients and clinicians), and treatment drop out. Secondary clinician outcomes include: extent of PracticeGround use with clients across clinicians' caseload.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* Meets DSM-IV criteria for MDD and/or DD
* Obtains a score of 11 or greater on the PHQ-9
* Currently receiving psychosocial treatment for depression by a study-participant clinician
* Payment-eligible to receive at least 12 weeks of additional psychosocial treatment

Exclusion Criteria:

* Current diagnosis of bipolar disorder or another psychotic disorder
* Active mania
* Current diagnosis of alcohol and/or drug dependence
* At imminent risk of suicide (as deemed by their clinician).

PROVIDERS

Inclusion Criteria:

* English speaker
* 18 years or older
* Currently licensed mental health treatment provider (or a therapist working towards licensure under direct supervision of licensed mental health treatment provider)
* Have an office with access to internet
* Have access to computer with sound card and/or tablet and printer
* Capacity to accept new patients seeking treatment for depressive symptoms

Exclusion Criteria:

* (PILOT ONLY) Receiving training for an evidence based treatment for depression, including behavioral activation, interpersonal therapy, cognitive/cognitive-behavioral therapy, mindfulness-based cognitive therapy or cognitive behavioral analysis system of psychotherapy
* Participated in the Field Test for WILLOW
* Is not comfortable/savvy with technology (by answering "I get easily frustrated and usually walk away from it" to the question "Which response best matches how you typically respond to complicated problems you encounter when using a new app, computer, or technology for the first time?"; answering "I am not comfortable and/or do not enjoy technology, particularly new forms of technology. I avoid the use of technology as much as is realistically possible." to the question "How technologically savvy/skilled are you?")
* Does not have a feasible office set up for using a computer in therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Evidence-Based Practice Institute, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited providers and their patients from 17 behavioral health clinics, outpatient clinics, and private practices. After consent, providers were randomized to WILLOW or TAU condition. Providers referred their existing new patients to the study; those deemed eligible and who consented were assigned to the same study condition as their provider.
Pre-assignment Details: 98 providers completed eligibility screening; 91 were eligible and 76 consented to participate. 29 participating providers enrolled 1+ patients. Providers referred 119 patients to the study; 100 completed screening, 73 met eligibility criteria, 66 provided consent, and 56 attended 4+ therapy sessions and completed all data collection points.
Groups:
- WILLOW: Clinicians have access to WILLOW's dynamic progress monitoring, clinical decision support, rich visual displays of client outcomes, online training modules in ESTs, just-in-time training for guided real-time assistance in delivering ESTs, educational videos, and a client portal.
  Evidence-based interventions for treating depression and concurrent problems in WILLOW included: Behavioral Activation for Depression, Cognitive Behavior Therapy for Insomnia, Collaborative Assessment and Management of Suicidality.
Period: Overall Study
Arm/Group | WILLOW | Treatment-as-Usual
Started | 80 (43 provider participants and 37 patient participants were assigned to the WILLOW condition.) | 62 (33 provider participants and 29 patient participants were assigned to the TAU condition.)
Completed | 49 (18 provider participants and 31 patient participants in the WILLOW condition completed participation) | 36 (11 provider participants and 25 patient participants in TAU condition completed study participation.)
Not Completed | 31 | 26
Not completed — No participating patient | 16 | 13
Not completed — Participant withdrew | 7 | 2
Not completed — Lost to Follow-up | 2 | 5
Not completed — Dropped/Excluded by PI | 6 | 6

BASELINE CHARACTERISTICS:
Population: Each participant completed baseline once. Provider participants who participated in both the pilot and the full RCT completed the baseline once overall rather than one in each study. 31 patient and 18 provider participants in the WILLOW condition; 25 patient and 11 provider participants in TAU were included were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | WILLOW | Treatment-as-Usual | Total
Number analyzed (Participants) | 49 | 36 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 35 | 83
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 43.4 [20 to 69] | 41.2 [18 to 79] | 42.5 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 25 | 16 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 38 | 28 | 66
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 49 | 36 | 85

OUTCOME MEASURES:

1. Primary Outcome: Depression, Anxiety, and Stress Scale (DASS)
Description: Higher scores on subscales from this 23-item measure reflected higher depression, anxiety, stress, and suicidality. Other researchers added two suicidality items to the original 21-item measure with permission from the original authors. Each subscale score is computed by summing the subscale items, then multiplying by 2. Total possible scores for the depression, anxiety, and stress subscales range from 0-42. We categorized DASS depression, anxiety, and stress scores into severity levels coded as 0, 1, and 2: Normal (0 through 9), Mild/moderate (10 through 20), and Severe/extremely severe (21 through 42) (Psychology Foundation of Australia, 2018). The DASS suicide subscale ranged from 0-12 and not recategorized.
Time Frame: baseline, 4 weeks, 8 weeks, 12 weeks
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WILLOW | Treatment-as-Usual
Number analyzed (Participants) | 31 | 25
score on a scale
  Baseline (depression subscale) | 1.55 (.68) | 1.68 (.56)
  Week 4 (depression subscale) | 1.32 (.79) | 1.4 (.65)
  Week 8 (depression subscale) | 1.1 (.75) | 1.08 (.76)
  Week 12 (depression subscale) | .94 (.94) | 1.08 (.76)
  Baseline (anxiety subscale) | .97 (.8) | .84 (.75)
  Week 4 (anxiety subscale) | .81 (.75) | .76 (.78)
  Week 8 (anxiety subscale) | .74 (.77) | .76 (.83)
  Week 12 (anxiety subscale) | .58 (.81) | .72 (.74)
  Baseline (stress subscale) | 1.55 (.68) | 1.60 (.58)
  Week 4 (stress subscale) | 1.32 (.70) | 1.16 (.69)
  Week 8 (stress subscale) | 1.29 (.64) | 1.24 (.72)
  Week 12 (stress subscale) | 1.10 (.75) | 1.00 (.76)
  Baseline (suicide subscale) | 3.42 (3.43) | 1.92 (2.68)
  Week 4 (suicide subscale) | 2.32 (3.31) | 1.28 (1.99)
  Week 8 (suicide subscale) | 1.68 (2.32) | 1.04 (1.84)
  Week 12 (suicide subscale) | 1.74 (3.26) | 1.52 (3.18)
Statistical Analysis 1: Comparison: WILLOW vs Treatment-as-Usual; We used the Generalized Linear Model to examine the between-condition change over time on study outcomes. We computed the design effects due to this nested design to determine the extent to which the intraclass correlation due to clustering and size of the cluster affected the analyses. Design effects ranged up to 1.8. Because all were under 2.0, we did not adjust analyses to account for clustering effects; Test type: Superiority; p = .734, Chi-squared — Analyses were performed on each subscale individually. This is the p-value for the Depression subscale; GEE Type III chi squared distribution with 3 degrees of freedom was used to examine between-condition change over time from baseline
Statistical Analysis 2: Comparison: WILLOW vs Treatment-as-Usual; We used a Generalized Linear Model to examine the between-condition change over time on study outcomes. We computed the design effects due to this nested design to determine the extent to which the intraclass correlation due to clustering and size of the cluster affected the analyses. Design effects ranged up to 1.8. Because all were under 2.0, we did not adjust analyses to account for clustering effects; Test type: Superiority; p = .27, Chi-squared — Analyses were performed on each subscale individually. This is the p-value for the Anxiety subscale; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: WILLOW vs Treatment-as-Usual; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .75, Chi-squared — Analyses were performed on each subscale individually. This is the p-value for the Stress subscale; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: WILLOW vs Treatment-as-Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .812, Chi-squared — Analyses were performed on each subscale individually. This is the p-value for the Suicide subscale; [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: Beck Depression Inventory (BDI-II)
Description: Higher scores on this 21-item reflect greater depressive symptoms in the past two weeks. All items are summed to a total score (possible range 0-63). We categorized BDI scores into severity levels coded as 0, 1, and 2: Minimal (raw scores 0 through 13), Mild/moderate (14 through 28), and Severe (29 through 63).
Time Frame: baseline, 4 weeks, 8 weeks, 12 weeks
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WILLOW | Treatment-as-Usual
Number analyzed (Participants) | 31 | 25
score on a scale
  Baseline | 1.25 (.63) | 1.52 (.65)
  Week 4 | 1.16 (.82) | 1.12 (.78)
  Week 8 | 1.00 (.78) | 1.08 (.76)
  Week 12 | .71 (.86) | 1.04 (.74)
Statistical Analysis 1: Comparison: WILLOW vs Treatment-as-Usual; We used the Generalized Linear Model to examine the between-condition change over time. We computed the design effects due to this nested design to determine the extent to which the intraclass correlation due to clustering and size of the cluster affected the analyses. Design effects ranged up to 1.8. Because all were under 2.0, we did not adjust analyses to account for clustering effects; Test type: Superiority; p = .036, Chi-squared; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: Higher scores on this ten-item measure reflects more severe depression. The total score (possible range 0-27) is created by summing the first nine items. We categorized PHQ severity levels coded as 0, 1, and 2 based on authors' research as minimal (0 through 4), mild/moderate (5 through 14), and moderately severe/severe (15 through 27). The recategorized scores are reported here.
Time Frame: baseline, 4 weeks, 8 weeks, 12 weeks
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WILLOW | Treatment-as-Usual
Number analyzed (Participants) | 31 | 25
score on a scale
  Baseline | 1.48 (.57) | 1.44 (.58)
  Week 4 | 1.23 (.62) | 1.24 (.60)
  Week 8 | 1.24 (.64) | 1.28 (.61)
  Week 12 | .97 (.71) | 1.08 (.76)
Statistical Analysis 1: Comparison: WILLOW vs Treatment-as-Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .664, Chi-squared; [statistical method as in outcome 1, analysis 1]

4. Primary Outcome: Behavioral Activation for Depression Scale Short Form (BADS-SF)
Description: The Behavioral Activation for depression Scale Short Form has 9 questions each having a scale from 0 (Not at All) to 6 (Completely) with a total range of 0-54. Higher scores on this nine-item scale reflect lower engagement in avoidance and higher engagement in activation behaviors over the course of BA for depression.
Time Frame: baseline, 4 weeks, 8 weeks, 12 weeks
Population: Patient Participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WILLOW | Treatment-as-Usual
Number analyzed (Participants) | 31 | 25
score on a scale
  Baseline | 18.8 (7.37) | 17.3 (6.47)
  Week 4 | 23.4 (9.42) | 20.4 (6.68)
  Week 8 | 24.6 (9.05) | 21.3 (7.52)
  Week 12 | 27.7 (8.42) | 23.6 (7.88)
Statistical Analysis 1: Comparison: WILLOW vs Treatment-as-Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .764, Chi-squared; [statistical method as in outcome 1, analysis 1]

5. Primary Outcome: Mental Health Services Satisfaction Survey (MHSSS)
Description: We created a ten-item measure in which higher scores reflected greater satisfaction with services they received. The measure had 10 questions each having a scale of 1(Strongly Disagree) to 5(Strongly Agree) with a total range of 10-50. Higher scores indicated a better outcome.
Time Frame: After first study therapy session, 4 weeks, 8 weeks, 12 weeks
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WILLOW | Treatment-as-Usual
Number analyzed (Participants) | 31 | 25
score on a scale
  Baseline | 37.6 (4.91) | 38.8 (7.24)
  Week 4 | 37.6 (6.77) | 37.8 (7.14)
  Week 8 | 39.2 (4.85) | 37.5 (9.00)
  Week 12 | 38.9 (7.14) | 38.3 (7.65)
Statistical Analysis 1: Comparison: WILLOW vs Treatment-as-Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .440, Chi-squared; [statistical method as in outcome 1, analysis 1]

6. Primary Outcome: Working Alliance Inventory (WAI)
Description: We modified this measure to include items from the BHS from Group Health. The resulting 12-item scale measures the therapeutic relationship with higher scores indicating stronger alliance. With 12 questions and each having a scale of 1(Never) to 7(Always) the total range was 12-84.
Time Frame: 4 weeks, 8 weeks, 12 weeks
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WILLOW | Treatment-as-Usual
Number analyzed (Participants) | 31 | 25
score on a scale
  Week 4 | 71.7 (10.44) | 71.9 (11.54)
  Week 8 | 73.7 (9.13) | 70.5 (11.23)
  Week 12 | 73.6 (10.46) | 72.7 (10.85)
Statistical Analysis 1: Comparison: WILLOW vs Treatment-as-Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .09, Chi-squared; GEE Type III chi squared distribution with 2 degrees of freedom was used to examine between-condition change over time

7. Primary Outcome: Therapy Task Checklist (TTC) - Patient Version
Description: We developed the TTC. The Therapy Task Checklist-Patient Version with 25 questions and each having a scale of 0 (Never/Very Rarely) to 7 (All of the Time) has a total range of 0-100. Higher scores reflected more frequent use of evidence-based therapy tasks, positive outcomes.
Time Frame: 4 weeks, 8 weeks, 12 weeks
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WILLOW | Treatment-as-Usual
Number analyzed (Participants) | 31 | 25
score on a scale
  Week 4 | 45.5 (18.76) | 37.9 (18.84)
  Week 8 | 46.6 (16.95) | 42.3 (19.48)
  Week 12 | 49.6 (19.70) | 39.0 (19.69)
Statistical Analysis 1: Comparison: WILLOW vs Treatment-as-Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .19, Chi-squared; GEE Type III chi squared distribution with 2 degrees of freedom was used to examine between-condition change over time from baseline

8. Primary Outcome: Modified Practice Attitudes Scale (MPAS)
Description: The Modified Practice Attitudes Scale with eight questions, each having a scale of 0 (Not at all) to 4(To a very great extent), has a total range of 0-32. Higher scores on this eight-item scale reflect more positive attitudes towards evidence-based practices.
Time Frame: Baseline, 12 weeks
Population: Provider participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WILLOW | Treatment-as-Usual
Number analyzed (Participants) | 25 | 23
score on a scale
  Baseline | 24.8 (3.06) | 24.9 (4.84)
  Week 12 | 24.6 (3.93) | 23.6 (5.77)
Statistical Analysis 1: Comparison: WILLOW vs Treatment-as-Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .15, Chi-squared; GEE Type III chi squared distribution with 1 degrees of freedom was used to examine between-condition change over time from baseline

9. Primary Outcome: Perceptions of Computer-Assisted Therapy Questionnaire (PCAT)
Description: The Perceptions of Computer-Assisted Therapy Questionnaire has 34 questions each having a scale of 1(Strongly Disagree) to 7 Strongly Agree). Thus, the total range was 34-238. Higher scores on this 34-item scale indicate stronger agreement with the benefits of computer-assisted therapy, or a better outcome.
Time Frame: Baseline, 12 weeks
Population: Provider participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WILLOW | Treatment-as-Usual
Number analyzed (Participants) | 25 | 23
score on a scale
  Baseline | 160.1 (19.39) | 157.4 (18.70)
  Week 12 | 170.4 (24.60) | 146.4 (21.70)
Statistical Analysis 1: Comparison: WILLOW vs Treatment-as-Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Chi-squared; [statistical method as in outcome 8, analysis 1]

10. Primary Outcome: ASA-Monitoring and Feedback Version (ASA-MF)
Description: The ASA-Monitoring and Feedback Version (ASA-MF) measure has 18 questions each having a scale of 1(Strongly Disagree) to 5(Strongly Agree) with a total range of 18-90. Higher scores on this 18-item scale reflect positive attitudes about standardized and routine progress monitoring, or positive outcomes.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Population: Provider participants. Sample sizes are smaller because this measure was e not used in the pilot study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WILLOW | Treatment-as-Usual
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 68.0 (6.24) | 64.8 (6.83)
  Week 4 | 72.1 (7.95) | 64.8 (6.47)
  Week 8 | 72.2 (7.56) | 68.3 (5.88)
  Week 12 | 71.1 (7.60) | 66.9 (3.90)
Statistical Analysis 1: Comparison: WILLOW vs Treatment-as-Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .14, Chi-squared; [statistical method as in outcome 1, analysis 1]

11. Primary Outcome: Monitoring and Feedback Attitudes Scale (MFA)
Description: The Monitoring and Feedback Attitudes Scale has 14 questions and each has a scale of 1(Strongly Disagree) to 5(Strongly Agree), thus the total range was 14-70. Higher scores on this 14-item measure indicate more positive attitudes about routine progress monitoring and providing feedback to patients about treatment progress, or positive outcomes.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Population: Provider participants. Sample sizes are smaller because the measure was not used in the pilot study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WILLOW | Treatment-as-Usual
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 57.9 (4.48) | 55.1 (5.68)
  Week 4 | 59.7 (5.67) | 57.2 (5.83)
  Week 8 | 58.9 (5.29) | 58.0 (6.71)
  Week 12 | 60.6 (5.88) | 60.1 (5.41)
Statistical Analysis 1: Comparison: WILLOW vs Treatment-as-Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .22, Chi-squared; [statistical method as in outcome 1, analysis 1]

12. Primary Outcome: Routine Monitoring (RM)
Description: We created a three-item measure where the total score is found by summing the items. The first two items are yes(scored 1)/no(scored 0) questions. The last item is a count measure that can be any number greater than or equal to 0. Thus, the total score can have any integer value greater than or equal to 0, with higher scores reflecting greater use of routine progress monitoring.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Population: Provider participants. Sample sizes are smaller because the measure was not used in the pilot study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WILLOW | Treatment-as-Usual
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 1.6 (1.76) | .60 (1.06)
  Week 4 | 4.6 (2.70) | 1.8 (1.36)
  Week 8 | 3.6 (2.39) | 1.3 (1.16)
  Week 12 | 3.3 (2.25) | 1.9 (1.36)
Statistical Analysis 1: Comparison: WILLOW vs Treatment-as-Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Chi-squared; [statistical method as in outcome 1, analysis 1]

13. Primary Outcome: Current Assessment Practice Evaluation-Revised (CAPER)
Description: We modified the original measure into nine items. The Current Assessment Practice Evaluation-Revised has 9 questions with each having a scale of 1(None, 0%) to 5 (Nearly All, 81-100%). Thus, the total range was 9-45 and higher scores reflect greater provider use of measurement-based care or positive outcomes.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Population: Provider participants. Sample sizes are smaller because the measure was not used in the pilot study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WILLOW | Treatment-as-Usual
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 17.6 (8.07) | 12.4 (5.04)
  Week 4 | 21.7 (9.66) | 13.2 (5.13)
  Week 8 | 21.9 (9.80) | 13.4 (5.66)
  Week 12 | 22.3 (11.26) | 13.4 (5.38)
Statistical Analysis 1: Comparison: WILLOW vs Treatment-as-Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .001, Chi-squared; [statistical method as in outcome 1, analysis 1]

14. Primary Outcome: Therapy Task Checklist (TTC) - Provider Version
Description: The Therapy Task Checklist -Provider Version has 22 questions and each have a scale of 0(Never/Very Rarely) to 4 (All of the time) with a total range of 0-88. Higher scores reflected more frequent use of evidence-based therapy tasks, or positive outcomes.
Time Frame: 4 weeks, 8 weeks, 12 weeks
Population: Provider participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WILLOW | Treatment-as-Usual
Number analyzed (Participants) | 25 | 23
score on a scale
  Week 4 | 48.7 (13.19) | 40.7 (12.51)
  Week 8 | 51.3 (13.33) | 43.7 (10.06)
  Week 12 | 50.8 (13.37) | 42.9 (7.91)
Statistical Analysis 1: Comparison: WILLOW vs Treatment-as-Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .99, Chi-squared; [statistical method as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data reporting was open throughout periods of recruitment and active participation of approximately 1 year and 8 months. It is noted that no adverse events were reported.
Description: PI's contact information were provided to participants in the consent form to self-report adverse outcomes (AE). Our Data Safety Monitoring Board (DSMB) did not anticipate AE stemming from the research because they identified it as a "protective study." In the event of an AE: PI notifies DSMB chair and IRB chair, DSMB chair determines whether to notify full DSMB, PI notifies IRB of the DSMB's recommended actions, and DSMB chair alerts NIMH Program Officer Adam Haim, PhD.
Arm/Group | WILLOW | Treatment-as-Usual
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/62
Other Adverse Events (participants affected / at risk) | 0/80 | 0/62

LIMITATIONS AND CAVEATS:
Overall study recruitment was lower than anticipated (target n=110). To address this, data from both pilot and full RCTs were included to maximize sample size and the Generalized Linear Model was used as it yields more power with missing data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT02314624/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT02314624/SAP_001.pdf
  • Informed Consent Form (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT02314624/ICF_002.pdf